CLINICAL TRIAL: NCT04875637
Title: Middle-ear Reflex Testing Using Wideband Acoustic Immittance
Acronym: WAI-MEMR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mimosa Acoustics (Industry)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WAI-MEMR-MA-16780-02
Record Dates: First submitted 2021-04-28; First posted 2021-05-06 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Hearing Disorders
Keywords: middle ear muscle reflex; wideband acoustic immittance
MeSH Terms: conditions — Hearing Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MEMR Diagnostic Evaluation (Other): Middle Ear Muscle Reflex using wideband acoustic reflectance to assess hearing status.
  Interventions: Diagnostic Test: WAI-MEMR

INTERVENTIONS:
Diagnostic Test: WAI-MEMR — Using wideband acoustic reflectance for middle-ear muscle reflex.

SUMMARY:
This project will assess the middle-ear muscle reflex using wideband acoustic immittance which is a valuable method for evaluating infants, children, and adults. The developments will facilitate clinical applications that include hearing screening and diagnostic evaluation of persons of all ages with normal hearing and with hearing loss.

DETAILED DESCRIPTION:
Measurement of middle-ear muscle reflexes (MEMR) constitutes an important component of the standard of care in auditory function assessment and diagnostic audiology. An important component of the middle-ear test battery involves characterizing neural function through the eighth nerve-brainstem pathway which is accomplished through measurement of the MEMR. The evaluation component of this project will involve testing of human subjects using wideband acoustic immittance in the evaluation of middle-ear muscle reflexes. Subjects in this project will be infants, children and adults with normal hearing as well as with conductive, sensory, and neural hearing loss. All subjects will receive wideband acoustic immittance (WAI) and middle-ear muscle reflex (MEMR) testing. Baseline testing includes pure tone audiometry and otoacoustic emissions.

ELIGIBILITY:
Inclusion Criteria:

* Normal hearing or hearing loss

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
WAI-MEMR | Through study completion, an average of 2 years
  MEMR threshold

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided